CLINICAL TRIAL: NCT05547919
Title: A Molecular Imaging-Derived Biomarker of PSMA Expression - Revealing Theranostic Potential in Gastroenterologic Tumors
Brief Title: PSMA in Gastroenterologic Tumors (GIPSMA)
Acronym: GIPSMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GI-PSMA22
Record Dates: First submitted 2022-08-26; First posted 2022-09-21 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastroenterologic tumors histologically positive for PSMA (Experimental): Tumor biopsy at baseline to establish diagnosis and to identify PSMA expression in an ex-vivo setting. Patients with ex-vivo PSMA expression receive a multimodal imaging approach: This includes a PSMA-targeted PET/CT (18F-PSMA) at baseline and conventional imaging.
  Interventions: Radiation: 18F-PSMA PET/CT

INTERVENTIONS:
Radiation: 18F-PSMA PET/CT — Patients with metastasized gastroenterologic tumors, that exhibit histological PSMA expression, receive an additional 18F-PSMA PET/CT to routine imaging.

SUMMARY:
The theranostic principle is based on the use of radiolabeled compounds which can be applied for diagnostic molecular imaging and targeted delivery of radiation to the tumor. Gastroenterologic tumors (GET), including hepatocellular Carcinoma, Colorectal Carcinoma, Pancreatic Adenocarcinoma, Cholangiocellular Carcinoma, gastroenteropancreatic neuroendocrine neoplasms also express a phenotypic biomarker called prostate-specific membrane antigen (PSMA), thereby rendering it a potential diagnostic (through positron emission tomography (PET) scan imaging) and therapeutic target for radioligand therapy. Aim is to evaluate whether PSMA-directed in-vivo imaging can be also applied to GET patients to determine if i) biopsy-derived tissue of newly diagnosed patients exhibit a PSMA expression profile, ii) PSMA-PET shows upregulated PSMA expression in-vivo, iii) such a molecular imaging approach identifies more disease sites relative to conventional imaging, and iv) if the PSMA PET signal predicts further clinical course and outcome under guideline-compatible treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed GET prior to initiation of guideline-compatible, anti-tumor therapy
* Available tissue specimen to conduct PSMA expression profiling
* Male/female, above 18 years old
* Patients must provide written informed consent
* Patients must be willing to comply with study procedures and available for follow-up examinations

Exclusion Criteria:

* Curative setting
* Not sufficient tumor tissue available
* Male Patients: No prostate carcinoma
* Other malignant neoplasms in patient's history
* Pregnancy or Breastfeeding
* Contraindications for PET/CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
True positive rate per patient specimen | 24 months
  The probability of GET is given when immunhistochemistry test is positive.
True positive rate per patient | 24 months
  The probability of GET is given when 18F-PSMA-1007 PET/CT is positive on a per patient basis.
Number of patients with identified tumor lesion sites | 24 months
  To compare the sites of disease identified on 18F-PSMA-1007 PET/CT in patients with GET to images derived by conventional imaging to evaluate the sensitivity of 18F-PSMA-1007 PET/CT.

SECONDARY OUTCOMES:
Ex-vivo PSMA expression | 24 months
  Expression of PSMA per specimen at immunhistochemistry.
PSMA uptake on 18F-PSMA-1007 PET | 24 months
  Quantified uptake of PSMA per tumor lesion basis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No